## Investigation of the Effects of Physiotherapy on Pain, Physical Function and Quality of Life in Patients with PRP Applied Knee Osteoarthritis

## Statistical methods used to compare groups

For descriptive statistics of quantitative variables; average, median, standard deviation, interquartile width will be given while for qualitative data; numbers and percentages will be used.

If the parameters provide normal distribution conditions, then parametric tests will be used for analysis. For the data to be considered significant, it will be desirable to be in the range of p < 0.05.

For intra-group and inter-group comparisons, the ANOVA test (in-between interactions) will be used which examines the intergroup and intergroup interaction. G-power software will be used to determine the power of statistical tests.